CLINICAL TRIAL: NCT01079364
Title: Better Acceptance of a Single Injection Apidra (Insulin Glulisine) Added to Once Daily Lantus (Insulin Glargine) Versus Twice Daily Premixed Insulin in a Real Life Use Setting
Brief Title: Better Acceptance of Single Injection Apidra Added to Once Daily Lantus Versus Twice Daily Premixed Insulin in Real Life Use Setting
Acronym: BASAAL PLUS
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Slow recruitment
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: APIDR_L_04717; 2009-015742-34 (EudraCT Number)
Record Dates: First submitted 2010-02-25; First posted 2010-03-03 (Estimated); Last update posted 2013-05-29 (Estimated); Status verified 2013-05

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — insulin glulisine; Insulin Glargine; insulin aspart, insulin aspart protamine drug combination 30:70

ARMS (2):
- Insulin glargine + Insulin glulisine (Experimental): Daily injection of insulin glargine plus one injection of mealtime insulin glulisine at the main meal
  Interventions: Drug: Insulin glulisine; Drug: Insulin glargine
- Premixed insulin (Active Comparator): twice daily premixed insulin (before breakfast and evening meal).
  Interventions: Drug: Premixed insulin (Insulin Aspart 30/70 )

INTERVENTIONS:
Drug: Insulin glulisine — Pharmaceutical form: boxes of 5 SoloStar® pens Route of administration: injection Dose regimen: once a day
  Other Names: Apidra®
  Arms: Insulin glargine + Insulin glulisine
Drug: Insulin glargine — Pharmaceutical form: boxes of 5 SoloStar® pens Route of administration: injection Dose regimen: once a day
  Other Names: Lantus®
  Arms: Insulin glargine + Insulin glulisine
Drug: Premixed insulin (Insulin Aspart 30/70 ) — Pharmaceutical form:boxes of 5 FlexPens Route of administration: Injection Dose regimen: twice daily
  Other Names: NovoMix 30/70®
  Arms: Premixed insulin

SUMMARY:
Primary Objective:

To demonstrate non-inferiority of once daily injection of insulin glargine (Lantus) plus one injection of mealtime insulin glulisine (Apidra) at the main meal versus twice daily premixed insulin (NovoMix 30/70) based on the reduction of HbA1c percentage from baseline to endpoint.

Secondary Objective:

* To determine treatment satisfaction (DTSQs/Diabetes Treatment Questionnaire - Status, DTSQc/ Diabetes Treatment Questionnaire - change and ITSQ/Insulin Treatment Satisfaction Questionnaire)
* To determine the mean HbA1c, FBG (Fasting Blood Glucose), prandial BG (Blood Glucose) and proportion of patients with a HbA1c <7%
* To determine the effect on adverse events (e.g. symptomatic hypoglycemic events, weight gain and injection site reactions)
* To determine the total insulin dose, average insulin glargine, insulin glulisine and premixed insulin dosages.

ELIGIBILITY:
Inclusion criteria:

* Patients with type 2 diabetes mellitus treated with insulin glargine once daily and oral blood glucose lowering medication
* Patients with a HbA1c > 7%
* Patients with a FBG within range (4-7 mmol/L) at baseline, based on the mean of 3 FBG values (measured 5x during the run-in phase, with the highest and lowest value excluded)

Exclusion criteria:

* Patients treated with an insulin other than insulin glargine
* Patients with hypersensitivity to insulin glargine, insulin glulisine, biphasic insulin aspart/insulin aspart protamine 30/70 or any of the excipients
* Patients with a (pre)proliferative retinopathy (an optic fundus examination should have been performed within the 2 years prior to study entry)
* Pregnant or lactating women
* Patients who are unable to fill in the PRO (Patient Reported Outcomes) questionnaires

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2010-01; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Glycosylated Haemoglobin (HbA1c) Value | at screening (week - 2), week 12 (if available) and 24
  Glycosylated Haemoglobin (HbA1c) is a biological parameter that reflects the blood glucose concentration over a long period of time. It is the standard parameter for glycemic control follow -up in diabetic patients.
Self Measured Blood Glucose (SMBG) | at Baseline (week 0), week 2, 12 and 24

SECONDARY OUTCOMES:
DTSQs (Diabetes Treatment Satisfaction Questionnaire - status) | at week 0, 12 and 24
DTSQc (Diabetes Treatment Satisfaction Questionnaire - change) | at week 24
ITSQ (Insulin Treatment Satisfaction Questionnaire) | at week 0, 12 and 24
Hypoglycemic events | at week 0, 2, 12 and 24
Adverse Events (excluding hypoglycemic events) | at week - 2, 0, 2, 12 and 24

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (1):
- Sanofi-Aventis Administrative Office, Gouda, Netherlands